CLINICAL TRIAL: NCT06840002
Title: An Open, Multicenter Phase Ib / II Clinical Study of SHR-A1811 Combined With Chemotherapy for Platinum Sensitive Recurrent Ovarian Cancer
Brief Title: A Clinical Study of SHR-A1811 Combined With Chemotherapy for Platinum Sensitive Recurrent Ovarian Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1811-216-OC
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-04

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Carboplatin; Bevacizumab; Oxaliplatin; Injections; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental)
  Interventions: Drug: SHR-A1811; Drug: Carboplatin; Drug: Bevacizumab; Drug: Oxaliplatin for Injection; Drug: Paclitaxel injection; Drug: Doxorubicin hydrochloride liposome injection; Drug: Adebrelimab Injection

INTERVENTIONS:
Drug: SHR-A1811 — SHR-A1811.
Drug: Carboplatin — Carboplatin.
Drug: Bevacizumab — Bevacizumab.
Drug: Oxaliplatin for Injection — Oxaliplatin for injection.
Drug: Paclitaxel injection — Paclitaxel injection.
Drug: Doxorubicin hydrochloride liposome injection — Doxorubicin hydrochloride liposome injetction.
Drug: Adebrelimab Injection — Adebrelimab injection.

SUMMARY:
The objective is to evaluate the tolerance, safety, pharmacokinetic characteristics and immunogenicity of SHR-A1811 combined with carboplatin and bevacizumab in the treatment of platinum sensitive recurrent epithelial ovarian cancer, and to determine the RP2D of the combination, and preliminarily to evaluate the effectiveness of SHR-A1811 combined regimen in the treatment of platinum sensitive recurrent epithelial ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily join this study, sign the informed consent form, have good compliance, and can cooperate with the follow-up.
2. Sufficient fresh or archived tumor tissue specimens can be provided for testing by the third-party central laboratory designated by the sponsor.
3. At least one measurable lesion conforming to RECIST v1.1.
4. ECOG PS score: 0-1.
5. Expected survival ≥ 12 weeks.
6. Female subjects with fertility must agree to comply with the contraceptive requirements from signing the informed consent form to 7 months after the last administration of the trial drug.

Exclusion Criteria:

1. With untreated or active central nervous system (CNS) tumor metastasis. Subjects with a history of meningeal metastasis or current meningeal metastasis.
2. Pleural effusion, pericardial effusion or peritoneal effusion with clinical symptoms, which cannot be well controlled.
3. Previous interstitial pneumonia or interstitial lung disease, non infectious pneumonia requiring steroid treatment.
4. With hypertension and cannot be well controlled by antihypertensive drug treatment.
5. Accompanied by poorly controlled or serious cardiovascular diseases.
6. Subjects with serious infection within 1 month before the first medication.
7. Have a history of immune deficiency, including HIV test positive, other acquired or congenital immune deficiency diseases, or a history of organ transplantation.
8. There are any other factors that may affect the results of the study or cause the forced termination of the study, such as alcohol abuse, drug abuse, criminal detention, and other serious diseases (including mental illness) that need combined treatment.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Dose limited toxicity (DLT) | Up to 21 days.
Recommended phase II dose (RP2D) | Up to 21 days.
Objective response rate (ORR) | Every 9 weeks lasting about one year.

SECONDARY OUTCOMES:
Duration of response (DoR) | Every 9 weeks lasting about one year.
Disease control rate (DCR) | Every 9 weeks lasting about one year.
Progression free survival (PFS) | Every 9 weeks lasting about one year.
Standard response rate (RR) | Every 9 weeks lasting about one year.
Overall survival (OS) | Approximately 3 years after the last subject enrolled.
Adverse events (AEs) | From the first drug administration to within 90 days after the last dose.
Serious adverse events (SAEs) | From the first drug administration to within 90 days after the last dose.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided